CLINICAL TRIAL: NCT00127738
Title: Renal Atherosclerotic Revascularization Evaluation: RAVE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 216-2004
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2006-02

CONDITIONS: Hypertension, Renovascular
Keywords: Hypertension; Renal artery stenosis; Kidney disease; Renal vascular disease; Atherosclerosis
MeSH Terms: conditions — Hypertension, Renovascular; Hypertension; Renal Artery Obstruction; Kidney Diseases; Atherosclerosis

INTERVENTIONS:
Procedure: Angiographic renal revascularization

SUMMARY:
The RAVE study will compare renal revascularization to medical management for people with atherosclerotic renal vascular disease (ARVD) and the indication for revascularization.

DETAILED DESCRIPTION:
It is uncertain whether patients with renal vascular disease will have renal or mortality benefits from re-establishing renal blood flow with renal revascularization procedures. Patients will be assessed for the standard nephrology research outcomes of progression to doubling of creatinine, need for dialysis, and death, as well as other cardiovascular outcomes. The investigators will also establish whether the use of a new inexpensive, simple and available ultrasound test, the renal resistance index (RRI), can identify patients with renal vascular disease who will not benefit from renal revascularization procedures.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg despite at least 3 antihypertensive medications
* Systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg on two antihypertensives with: a rise in creatinine > 20% after initiation of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB); the sudden onset of hypertension occurring after age 55; hypokalemia or the presence of an abdominal bruit; a history of flash pulmonary edema; or any three of: peripheral vascular disease, coronary artery disease, cerebrovascular disease, smoking, hyperlipidemia, diabetes or male gender.

Exclusion Criteria:

* Serum creatinine > 220 umol/L or estimated glomerular filtration rate (GFR) by Cockroft-Gault equation < 20 ml/min
* Patients who are unwilling or unable to give informed consent
* Known contraindication to renal revascularization such as anaphylactic allergy to contrast dye
* An abdominal aortic aneurysm requiring surgery
* A single functioning kidney; a total occlusion of the renal artery or renal artery stenosis due to fibromuscular dysplasia.
* Previous revascularization

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-01; Study Completion 2006-12

PRIMARY OUTCOMES:
Dialysis
Death
Doubling of creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Tobe, MD, Principal Investigator — Sunnybrook & Women's College Health Sciences Centre
Locations (1):
- Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tobe SW, Atri M, Perkins N, Pugash R, Bell CM. Renal athersosclerotic revascularization evaluation (RAVE study): study protocol of a randomized trial [NCT00127738]. BMC Nephrol. 2007 Jan 26;8:4. doi: 10.1186/1471-2369-8-4. PMID 17257413